CLINICAL TRIAL: NCT04421859
Title: Augmented Reality Mobile Application for Glaucoma Education in the South Bronx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx-Lebanon Hospital Center Health Care System (Other)
Collaborators: EyeCU Group (Unknown); VISRE (Unknown)
Responsible Party: Principal Investigator, Dr. Stephen Lau, Ophthalmology Resident, Bronx-Lebanon Hospital Center Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11141902
Record Dates: First submitted 2020-05-29; First posted 2020-06-09 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EyeCU App (Experimental): Augmented reality mobile application called "EyeCU" which simulates glaucoma progression and enhances understanding about the disease and its course. It is a bilingual (English/Spanish) application that is free-to-download on the Android and Apple app store. It will be delivered on a hospital owned tablet device and patients will be instructed to complete two sections, taking approximately 10 minutes.
  Interventions: Other: EyeCU Mobile Application

INTERVENTIONS:
Other: EyeCU Mobile Application — Augmented reality glaucoma education mobile phone application

SUMMARY:
A team at the National Healthcare Group Eye Institute in Singapore have developed an augmented reality mobile phone application, EyeCU, to simulate glaucoma progression and enhance understanding about the disease and its course. It is a bilingual (English/Spanish) application that is free-to-download on the Android and Apple app store. As eye care physicians in the South Bronx, the investigators are hopeful that the findings in this study can be extrapolated to our patients in the South Bronx, where poor health literacy, non-adherence to glaucoma medication and poor follow-up remains a large barrier. The investigators hope that by offering the simulation in both English and Spanish, the investigators will not only be able to improve our patients' understanding of glaucoma, but also improve glaucoma treatment adherence and assess our patient population's responsiveness to augmented reality as an educational platform.

DETAILED DESCRIPTION:
Experimental design: Pilot cohort study

Data collection: Patient characteristics such as age, sex, ethnicity, preferred language, zip code, employment status, highest educational attainment, current topical eye medications, Past Ocular History, Past Medical History

Recruitment for participation in the study will be performed during glaucoma clinic registration Consent will be conducted by a member of the research team who is not directly involved in the participant's clinical care Pre-intervention glaucoma knowledge questionnaire (NEHEP glaucoma knowledge questionnaire) will be given to participants, to be completed on dedicated clinic tablet device.

Post-intervention glaucoma knowledge questionnaire (NEHEP glaucoma knowledge questionnaire) will be given to participants, to be completed on dedicated clinic tablet device.

Rate of missed glaucoma follow-up appointments before and 6 months after application use will be collected from the electronic medical record.

Rate of medication adherence before and 6 months after application use will be collected from the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a clinical diagnosis of glaucoma on medical therapy for at least 4 months

Exclusion Criteria:

* Patients with optic neuropathies unrelated to glaucoma
* Patients with VA 20/100 or worse in both eyes
* Visual defects involving fixation in both eyes
* Patients with symptoms impairing ability to operate a smartphone during visit including diplopia, motor difficulties, cognitive impairment, illiteracy
* Patients who are unable to read or understand English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Questionnaire Scores | From date of intervention to date of post-intervention NEHEP glaucoma knowledge test, assessed up to 2 months
  Scores of pre- and post-intervention NEHEP glaucoma knowledge questionnaires will be compared
Change in Follow Up Adherence | Before and 6 months after intervention
  Attendance rate at glaucoma follow-ups will be collected from electronic medical record
Change in Medication Adherence | Before and 6 months after intervention
  Self-reported adherence to glaucoma medications will be collected from electronic medical record

CONTACTS AND LOCATIONS:
Locations (1):
- BronxCare Health System, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No